CLINICAL TRIAL: NCT04138368
Title: The Effect of Early Dyadic Psychotherapeutic Intervention for Mothers Suffering From PPD on Oxytocin Level and on Childrens' Emotional and Behavioral Development
Brief Title: The Effect of Early Dyadic Psychotherapy for Mothers Suffering From PPD on Oxytocin Level and on Childrens' Emotional Development
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Guy Schusheim, Director of child and Adolescent Outpatient Psychiatric Clinic, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EMC-0057-19
Record Dates: First submitted 2019-09-26; First posted 2019-10-24 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dyadic treatment (Experimental): Mothers and infants will be treated with dyadic psychotherapy focused on interactions, emphasizing eye contact, body language, empathy, and social reciprocity, using the principles of Interaction Guidance Therapy (Sameroff et al., 2004). Dyadic psychotherapy will be administered one time a week during the 8-week trial period, at the subject's home. Each session, approximately 90 minutes long, will include videotaping mother-infant interaction, watching the last session's interaction as a part of video-feedback technique, and discussing main issues in the mother-infant relationship. In addition, each session will begin and end with a- 5-minute episode of affectionate touch and gaze synchrony between the mother and her infant.
  Interventions: Behavioral: dyadic psychotherapeutic intervention
- supportive treatment (Active Comparator): mothers will receive psychoeducational knowledge regarding the infants' development. The treatment will be administered one time a week during the 8-week trial period, at the subjects' home.
  Interventions: Behavioral: supportive intervention

INTERVENTIONS:
Behavioral: dyadic psychotherapeutic intervention — Mothers and infants will be treated with dyadic psychotherapy focused on interactions, emphasizing eye contact, body language, empathy, and social reciprocity, using the principles of Interaction Guidance Therapy (Sameroff et al., 2004). Dyadic psychotherapy will be administered one time a week during the 8-week trial period, at the subject's home. Each session, approximately 90 minutes long, will include videotaping mother-infant interaction, watching the last session's interaction as a part of video-feedback technique, and discussing main issues in the mother-infant relationship. In addition, each session will begin and end with a- 5-minute episode of affectionate touch and gaze synchrony between the mother and her infant.
  Arms: dyadic treatment
Behavioral: supportive intervention — Supportive therapy: mothers will receive psychoeducational knowledge regarding the infants' development. The treatment will be administered one time a week during the 8-week trial period, at the subjects' home.
  Arms: supportive treatment

SUMMARY:
Background: Postpartum depression follows approximately 10-15% of deliveries. Maternal functional disability, particularly in the relationship with the infant, a hallmark of PPD, causes impairment in the mother's ability to bond with her infant. Subsequently, this impairment leads to deleterious long-term consequences for infant cognitive, neurological, and social-emotional growth, and is associated with psychiatric disorders in later life. Therefore, the development of effective short-term treatment in such a highly prevalent phenomenon is of a high clinical priority. While pharmacological and psychological treatments are effective in treating PPD , these interventions have failed to show a significant improvement in mother-child interaction quality and infant development.

The Oxytocin System: Oxytocin (OXT) is a nine amino acid neuro-peptide, found exclusively in mammals and is released during labor and lactation. Among the central influences of OXT on human social behavior are increased trust, empathy and eye contact. Brain imaging found that maternal attachment activates regions in the brain's reward systems that are rich with oxytocin and vasopressin receptors . Such findings led researchers to speculate that OXT may be involved in linking and maintaining the connection between social recognition systems and feelings of pleasure . According to this speculation, pair bonding is a form of conditioned reward learning, whereby OXT promotes the reward in social encounters, thus enhancing the motivation to engage in such interaction .

Disruptions to the oxytocin system in depression have been repeatedly observed, and woman suffering from PPD have lower plasma OXT concentrations in comparison to the control group . A recent small treatment study of OXT in women suffering from PPD did not show a positive effect on mood; however, it did show improved mother-child interactions.

Studies suggest a bio-behavioral feedback loop of OXT, parenting, and infant social competence. Rationale and Hypotheses of the Current Research: We speculate that mothers suffering from PPD exhibit high levels of depression and low levels of OXT, hence experiencing the interaction with their child as less rewarding, which in turn promote further depressive symptoms and interfere with child development.

The aims of this study are:

1. To assess the relationship between levels of oxytocin in mothers suffering from postpartum depression and their babies, before and after psychological dyadic treatment compered to supportive treatment.
2. To study the added value of dyadic treatment over conventional supportive treatment for PPD that does not focus specifically on the mother's relationship with her baby.
3. To show the effects of dyadic treatment for PPD mothers and their children on the child's emotional and behavioral development.

Methods: Subjects: 50 Mothers will be interviewed and diagnosed as suffering from PPD according to DSM-IV-TR, will be enrolled within 2-8 months postpartum.

DETAILED DESCRIPTION:
Background: Postpartum depression follows approximately 10-15% of deliveries. Maternal functional disability, particularly in the relationship with the infant, a hallmark of PPD, causes impairment in the mother's ability to bond with her infant. Subsequently, this impairment leads to deleterious long-term consequences for infant cognitive, neurological, and social-emotional growth, and is associated with psychiatric disorders in later life. Recently, biological correlates of maternal deprivation and maternal depression on the infant's brain in both animal and human studies have been found . Therefore, the development of effective short-term treatment in such a highly prevalent phenomenon is of a high clinical priority. While pharmacological and psychological treatments are effective in treating PPD, these interventions have failed to show a significant improvement in mother-child interaction quality and infant development.

The Oxytocin System: Oxytocin (OXT) is a nine amino acid neuro-peptide, found exclusively in mammals and is released during labor and lactation. The effects of OXT on the anterior cingulate, OFC and vmPFC, suggesting its effect on 'social brain' areas have been reported in the past , including modulation of maternal behaviors and paternal behaviors including positive affect, social gaze, touch, and vocal synchrony with the infant . Among the central influences of OXT on human social behavior are increased trust , empathy and eye contact . Brain imaging found that maternal attachment activates regions in the brain's reward systems that are rich with oxytocin and vasopressin receptors . Such findings led researchers to speculate that OXT may be involved in linking and maintaining the connection between social recognition systems and feelings of pleasure . According to this speculation, pair bonding is a form of conditioned reward learning, whereby OXT promotes the reward in social encounters, thus enhancing the motivation to engage in such interaction .

Disruptions to the oxytocin system in depression have been repeatedly observed, and woman suffering from PPD have lower plasma OXT concentrations in comparison to the control group . Recent studies investigated the therapeutic potential of OXT in psychopathologies involving impaired social functioning such as autism spectrum disorders where OXT was found to facilitate social information processing and retention of social information, in social anxiety disorder , and schizophrenia where OXT administration resulted in a significant improvement in several social cognition measures and symptom reduction. Furthermore, a recent small treatment study of OXT in women suffering from PPD did not show a positive effect on mood; however, it did show improved mother-child interactions.

Studies suggest a bio-behavioral feedback loop of OXT, parenting, and infant social competence. The mechanisms of cross-generation transmission in the OXT system have been observed in human parents and infants in the first months of the infant's life and showed that parent and child's OXT levels are highly correlated and higher parental OXT was associated with higher infant OXT. Studies in non-human primates have shown long-term consequences on the development of social competence and infant's ultimate parental skills.

Rationale and Hypotheses of the Current Research: We speculate that mothers suffering from PPD exhibit high levels of depression and low levels of OXT, hence experiencing the interaction with their child as less rewarding, which in turn promote further depressive symptoms and interfere with child development.

The aims of this study are:

1. To assess the relationship between levels of oxytocin in mothers suffering from postpartum depression and their babies, before and after psychological dyadic treatment compered to supportive treatment.
2. To study the added value of dyadic treatment over conventional supportive treatment for PPD that does not focus specifically on the mother's relationship with her baby.
3. To show the effects of dyadic treatment for PPD mothers and their children on the child's emotional and behavioral development.

Methods: Subjects: 50 Mothers will be interviewed and diagnosed as suffering from PPD according to DSM-IV-TR, will be enrolled within 2-8 months postpartum.

Procedure:

An informed consent will be obtained, inclusion and exclusion criteria will be examined, demographic information, psychiatric and medical history will be obtained, and MADRS, CGI-S, and GAD7 questionnaires will be performed.

The baseline assessment will be conducted at the infant's home, at that time, a mother -infant interaction will be videotaped, and the YIPTA, BDI, EPDS, STAI, PSI, NMR, ERC, IOS, PBI, EQ and IRI questionnaires will be administered. Salivary OXT samples will be collected from the infants and salivary OXTsamples will be collected from the parent .

Women with PPD will be invited for a mid-point clinical evaluation at the outpatient Psychiatric Department, Haemek Medical Center. The evaluation will include a psychiatric evaluation using MADRS, CGI-S, and GAD-7 questionnaires.

the women in the PPD group will participate in 8 weeks of dyadic psychotherapy (DP) combining video feedback. The treatment will be conducted at the subject's home. Additional 25 PPD women will receive only supportive treatment at their home. The supportive treatment will include psychoeducation regarding the development of the infant. During the 8-week treatment, salivary OXT,Estradiol, Progesterone, SIGA and Vasopressin samples will be collected from the mother and infant at the beginning and the end of each session.

Four weeks into DP, women with PPD will undergo another clinical evaluation at the outpatient Psychiatric Department, Haemek Medical Center.

A final end-of-study clinical evaluation, for all women in the groups, will be conducted at the end of 12 weeks. Another assessment will be conducted at the infant's home, including mother -infant interaction. Mother-infant interaction will be filmed and assessed using the CIB Manual and the NOLDOS coding system. Salivary OXT, Estradiol, Progesterone, SIGA and Vasopressin samples will be collected from the mother and from the infant. PPD and control mothers. For PPD mothers, the evaluation will include a psychiatric evaluation (MADRS, CGI-S, and GAD-7 the MADRS) and the emotional conflict task at the outpatient Psychiatric Department, Haemek Medical Center.

Study duration: The study is expected to proceed for approximately 2 years. First year: setting up study infrastructure, preparation of collaborations, beginning of patient recruitment and treatment. Second year: patient recruitment and treatment according to protocol and data analysis.

ELIGIBILITY:
Inclusion Criteria:

* women age 18 years old +
* women screening score of Depression EPDS>10 (Edinburgh quastionnnaire)
* single child delivery
* babies 3-8 monthes years old

Exclusion Criteria:

* severe MDD
* intelectual disability
* women screening score of Depression EPDS<10 (Edinburgh quastionnnaire)
* pregnant women
* women diagnosed with Bipolar disorder or Schizophrenia, delirium, psychosis *due to drug abuse, OCD
* Aggressive intentions towards the baby
* high risk for self and other injury
* drug abuse
* physical condition influencing depressive symptoms
* unstable physical condition due to various illnesses (cancer, diabetes...)

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
the dyadic psychotherapy reinforce mother-child bonding and attachment, over and above the standard supportive care. | 8 weeks of treatment
  Oxytocin levels under dyadic therapy will be higher compared to the control group
the dyadic psychotherapy will prevent the development of emotional psychopathology of the child | 18 monthes of life
  Dyadic therapy will reduce behavioral and developmental problems

CONTACTS AND LOCATIONS:
Locations (1):
- Ilanir shchori, Afula, Israel

IPD SHARING:
Plan to Share IPD: No